CLINICAL TRIAL: NCT07054619
Title: The Effect of Experiential Learning Based First Aid Training on Knowledge and Self-Sufficiency of Parents of Intellectual Disability Children: A Randomized Controlled Trial
Brief Title: How First Aid Training Helps Parents of Children With Intellectual Disabilities
Acronym: ELFAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Ayse Sezer Balci, Assistant Professor of Nursing, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GO=2022/522
Record Dates: First submitted 2025-06-02; First posted 2025-07-08 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Intellectual Disability, Mild; First Aid Training
Keywords: First Aid Training Experiential Learning Intellectual Disability Parental Education Randomized Controlled Trial Self-Sufficiency
MeSH Terms: conditions — Intellectual Disability; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Control Group (No Intervention): Participants in this group did not receive any training during the study but were provided with printed first-aid educational materials after completing the post-test.
- Experimental: Training Group (Experimental): Participants received four sessions of first-aid training based on Kolb's Experiential Learning Model, including real-life simulations and group exercises.
  Interventions: Behavioral: Experiential First Aid Training

INTERVENTIONS:
Behavioral: Experiential First Aid Training — A first aid training program based on Kolb's Experiential Learning Model conducted in four sessions using real-life scenarios and group exercises.
  Arms: Experimental: Training Group

SUMMARY:
itle: How First Aid Training Helps Parents of Children With Intellectual Disabilities

Purpose:

This study aims to find out how experiential learning-based first aid training affects the knowledge and self-sufficiency of parents who have children with intellectual disabilities.

Who Can Participate:

Parents of children with intellectual disabilities are invited to take part in this study.

What Happens During the Study:

Participants will attend a first aid training program based on experiential learning. Their knowledge and ability to care for their children will be measured before and after the training.

Risks and Benefits:

There are no significant risks involved. Parents may benefit by gaining important first aid skills, which can help them better protect and support their children.

Contact Information:

If you have any questions or want to learn more about the study, please contact [asbalci@mehmetakif.edu.tr].

DETAILED DESCRIPTION:
This study investigates how first aid training based on experiential learning affects the knowledge and self-sufficiency of parents with children who have intellectual disabilities. The research is designed as a randomized controlled trial, which means participants will be randomly assigned to either the intervention group receiving the training or a control group that does not.

The experiential learning approach involves hands-on activities, simulations, and interactive sessions aimed at improving the parents' practical first aid skills. The study will measure changes in parents' knowledge and confidence in providing first aid before and after the training.

The outcomes of this research will help determine whether this type of training can empower parents to better respond to emergencies involving their children, potentially improving safety and wellbeing.

ELIGIBILITY:
Inclusion Criteria

* Parents of children diagnosed with intellectual disabilities
* Age of parents: 18 years and older
* Willingness to participate in first aid training
* Able to communicate in the language of the training

Exclusion Criteria

* Received formal first-aid training within the last 12 months
* Cognitive impairments preventing comprehension of training content
* Unwilling or unable to attend all training sessions and assessments

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Change in First-Aid Knowledge Score (pre- and post-training) | Baseline and immediately post-intervention
  First Aid Knowledge Questionnaire (self-developed; score range: 0-20; higher scores indicate better knowledge)
Change in First-Aid Self-Efficacy Score | Baseline and immediately post-intervention
  Home Accidents First Aid Self-Efficacy Scale (score range: 10-50; higher scores indicate greater self-efficacy)

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy University Faculty of Health Science, Burdur, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (e.g., demographic data, first-aid knowledge scores, self-efficacy scores) will be shared with qualified researchers upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Within 6 months of publication, available for 5 years
Access Criteria: Data will be shared upon request via email to the principal investigator.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT07054619/Prot_SAP_001.pdf